CLINICAL TRIAL: NCT06141369
Title: Treatment of Advanced Endocrine Tumor With Iindividualized mRNA Neoantigen Vaccine (mRNA-0523-L001)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Guang Ning, Principal Investigator, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2023-161
Record Dates: First submitted 2023-11-13; First posted 2023-11-21 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Adrenal Cortical Carcinoma; Medullary Thyroid Cancer; Thymic Neuroendocrine Carcinoma; Pancreatic Neuroendocrine Tumor
MeSH Terms: conditions — Adrenocortical Carcinoma; Carcinoma, Medullary; Adenoma, Islet Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mRNA-0523-L001 (Experimental): individualized mRNA neoantigen vaccine (mRNA-0523-L001)
  Interventions: Biological: individualized mRNA neoantigen vaccine (mRNA-0523-L001)

INTERVENTIONS:
Biological: individualized mRNA neoantigen vaccine (mRNA-0523-L001) — Individualized mRNA neoantigen vaccine (mRNA-0523-L001) will be injected intramuscularly every 21 days for 9 cycles. Dose escalation will be administered in 3 patients. 18 additional patients will be recruited and administered at the maximum tolerated(MTD) dose for all nine cycles.

SUMMARY:
Treatment of advanced endocrine tumors, including adrenal corticocarcnioma (ACC), medullary thyroid carcinoma (MTC), thymic neuroendocrine tumor and pancreatic neuroendocrine tumor is challenging. Previous genomic profiling studies showed they presented a number of somatic mutations. The tumors Individualized mRNA neoantigen vaccine provide a promising solution since a significant portion of these tumors showed high quality of tumor specific neoantigen. The primary objective is to observe and evaluate the safety and tolerability of individualized mRNA neoantigen vaccine (mRNA-0523-L001) for the treatment of advanced endocrine tumors, failure of standard treatment or no standard treatment currently available. The secondary objective is to observe the preliminary efficacy of mRNA-0523-L001 for the treatment of advanced endocrine tumors, failure of standard treatment or no standard treatment currently available, including:

1. Neoantigen-specific CD4+ and CD8+ T lymphocyte responses induced by mRNA-0523-L001;
2. Objective response rate (ORR) and disease control rate (DCR) of tumors;
3. Progression-free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily sign the written informed consent form and can comply with the visits and related procedures specified in the protocol;
2. The subjects are 18 years old or older, regardless of gender;
3. Patients with advanced endocrine tumors confirmed by histology or cytology in the past 6 months (including medullary thyroid carcinoma, thymic carcinoma and adrenal cortical carcinoma, etc.), who have failed standard treatment or have no standard treatment available;
4. No HLA-related genes or chromosomal regions with copy number variations (CNVs) or loss of heterozygosity (LOH) were detected by gene sequencing;
5. They have advanced or metastatic lesions confirmed by immunohistochemistry, and have frozen tissue/cells sufficient for WES and RNAseq sequencing, and after bioinformatics analysis, they predict at least one antigen that is effectively presented by their own HLA, such as KRAS or TP53 mutations and corresponding HLA typing, see 1.4 for the rationale of the topic.
6. Expected survival ≥ 4 months;
7. According to the Response Evaluation Criteria in Solid Tumors (RECIST 1.1), they have at least one measurable lesion, which should not have received local treatment such as radiotherapy (lesions in the previous radiotherapy area, if confirmed to have progressed, can also be selected as target lesions);
8. Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0 or 1;
9. They have not used granulocyte colony-stimulating factor (G-CSF), granulocyte-macrophage colony-stimulating factor (GM-CSF), red blood cell transfusion or platelet transfusion within 14 days before the examination.
10. Subjects of childbearing potential (male and female) who meet the inclusion criteria must agree to use reliable contraception methods (hormonal or barrier methods or abstinence) during the trial and for at least 90 days after the last administration; women of childbearing age must have a negative blood pregnancy test within 7 days before the first administration.
11. Virology test: No CMV, EBV, HIV, HBV, HCV, syphilis infection (only at baseline)

Exclusion Criteria:

1. Received chemotherapy, hormone therapy, traditional Chinese medicine with anti-tumor indications or other anti-tumor treatments within 4 weeks before the first administration (for mitomycin and nitrosourea, the last administration was within 6 weeks before the first administration of this study drug), or within 5 half-lives of immunotherapy or molecular targeted therapy;
2. Received other major surgery other than diagnosis or biopsy within 4 weeks before the first administration, or expected to receive major surgery during the study;
3. Patients who have received allogeneic hematopoietic stem cell transplantation or organ transplantation in the past, or plan to receive organ transplantation during this study;
4. Patients who have received other tumor vaccines or cell therapies in the past; Medical condition
5. Patients with clinically symptomatic brain metastases, spinal cord compression, carcinomatous meningitis, or other evidence indicating that the patient's brain or spinal cord metastases are not controlled, and are deemed unsuitable for enrollment by the investigator;
6. In the past 2 years, there have been known other malignant tumors that are progressing or require active treatment (except for non-melanoma skin cancer, superficial bladder cancer, and cervical carcinoma in situ that have been cured by radical surgery);
7. Have a history of interstitial lung disease (ILD) or pulmonary interstitial fibrosis;
8. Have a history of severe cardiovascular and cerebrovascular diseases, including but not limited to: a) Have severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias requiring clinical intervention, II-III degree atrioventricular block; corrected QTc interval male > 450 milliseconds, female > 470 milliseconds, b) Acute coronary syndrome, congestive heart failure, aortic dissection, stroke or other grade 3 or higher cardiovascular and cerebrovascular events occurred within 6 months before the first administration, c) New York Heart Association (NYHA) ≥ III grade heart failure or left ventricular ejection fraction (LVEF) <50%.
9. Other serious and/or uncontrollable diseases that may affect the subject's participation in this study, as determined by the investigator, including but not limited to: a) Have a history of severe drug allergy, or known to be allergic to any component of the tumor vaccine; or have had a severe allergic reaction to other monoclonal antibodies in the past, b) Have a history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases, c) Evidence of severe or uncontrolled liver or kidney disease, d) Poorly controlled hypertension, diabetes, etc., e) Patients with active ulcers or gastrointestinal bleeding f) Have a severe infection that requires intravenous infusion of antibiotics or hospitalization; or uncontrolled active infection within 4 weeks before the first administration, g) Have active syphilis infection.
10. Participated in other clinical trials within 4 weeks before the first administration (except for screening failure);
11. Currently receiving systemic use of corticosteroids (except for recent or current use of inhaled corticosteroids);
12. Pregnant or lactating women; Laboratory and imaging examinations
13. Imaging (CT or MRI) shows that the tumor invades the large blood vessels and has a tendency to bleed;
14. Have clinically significant thyroid function abnormalities, and the investigator deems them unsuitable for enrollment;
15. Active pneumonia was found in the screening chest CT scan;
16. Uncontrolled pleural effusion, pericardial effusion, or ascites that requires repeated drainage;
17. The adverse reactions of previous anti-tumor treatment have not recovered to NCI-CTCAE 5.0 grade evaluation ≤ 1 (except for hair loss);
18. Hepatitis B surface antigen (HBsAg) positive and peripheral blood hepatitis B virus deoxyribonucleic acid (HBV DNA) test value higher than the upper limit of normal; hepatitis C virus antibody (HCV Ab) positive and HCV RNA test value higher than the upper limit of normal; Investigator assessment
19. The investigator considers that there are other reasons that are not suitable for participating in the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-01-13 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) or Dose-limiting toxicity (DLT).If MTD is not reached, Biologically Effective Dose (BED)tumor neoantigen. | At the end of cycle 1(each cycle is 21 days)
  The highest dose of a drug or treatment that does not cause unacceptable side effects.
Incidence of treatment-related adverse events. | At the end of cycle 1(each cycle is 21 days)
  According to National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE v5.0).

SECONDARY OUTCOMES:
Reaction of antigen-specific T cells in peripheral blood. | At the end of cycle 1(each cycle is 21 days)
  mRNA-0523-L001 personalized tumor vaccine induces neoantigen specific CD4+and CD8+T lymphocyte responses.
Objective tumor response rate (ORR) | At the end of cycle 1(each cycle is 21 days)
  ORR calculates the ratio of the number of patients whose best response is complete remission (CR) or partial remission (PR) to the total number of evaluable patients according to RECIST 1.1 criteria. Those who have not been evaluated for lesion and tumor response will be regarded as non-evaluable patients and will not be counted.
Disease control rate (DCR) | At the end of cycle 1(each cycle is 21 days)
  DCR calculates the ratio of the number of patients whose best response is complete remission (CR), or partial remission (PR), or stable disease (SD) to the total number of evaluable patients according to RECIST 1.1 criteria. Those who have not been evaluated for lesion and tumor response will be regarded as non-evaluable patients and will not be counted.
Progressive free survival (PFS) | At the end of cycle 1(each cycle is 21 days)
  Progression-free Survival of Personalized mRNA Tumor Vaccine.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin hospital, Shanghai Jiao-Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hofland J, Kaltsas G, de Herder WW. Advances in the Diagnosis and Management of Well-Differentiated Neuroendocrine Neoplasms. Endocr Rev. 2020 Apr 1;41(2):371-403. doi: 10.1210/endrev/bnz004. PMID 31555796
- [Background] Saltiki K, Simeakis G, Karapanou O, Alevizaki M. MANAGEMENT OF ENDOCRINE DISEASE: Medullary thyroid cancer: from molecular biology and therapeutic pitfalls to future targeted treatment perspectives. Eur J Endocrinol. 2022 Jul 26;187(3):R53-R63. doi: 10.1530/EJE-22-0312. Print 2022 Sep 1. PMID 35895692
- [Background] Fazzari F, Mantovani R, Donghi V, Curzi M, Bragato RM. From EACVI recommendations to the real-world experience: safety of performing echocardiography in the pandemic era. Eur Heart J Cardiovasc Imaging. 2021 Jun 22;22(7):e82-e83. doi: 10.1093/ehjci/jeab010. No abstract available. PMID 33491077
- [Background] Ciampi R, Romei C, Ramone T, Prete A, Tacito A, Cappagli V, Bottici V, Viola D, Torregrossa L, Ugolini C, Basolo F, Elisei R. Genetic Landscape of Somatic Mutations in a Large Cohort of Sporadic Medullary Thyroid Carcinomas Studied by Next-Generation Targeted Sequencing. iScience. 2019 Oct 25;20:324-336. doi: 10.1016/j.isci.2019.09.030. Epub 2019 Sep 26. PMID 31605946
- [Background] Tran E, Robbins PF, Rosenberg SA. 'Final common pathway' of human cancer immunotherapy: targeting random somatic mutations. Nat Immunol. 2017 Feb 15;18(3):255-262. doi: 10.1038/ni.3682. PMID 28198830
- [Background] Parikh AR, Mojtahed A, Schneider JL, Kanter K, Van Seventer EE, Fetter IJ, Thabet A, Fish MG, Teshome B, Fosbenner K, Nadres B, Shahzade HA, Allen JN, Blaszkowsky LS, Ryan DP, Giantonio B, Goyal L, Nipp RD, Roeland E, Weekes CD, Wo JY, Zhu AX, Dias-Santagata D, Iafrate AJ, Lennerz JK, Hong TS, Siravegna G, Horick N, Clark JW, Corcoran RB. Serial ctDNA Monitoring to Predict Response to Systemic Therapy in Metastatic Gastrointestinal Cancers. Clin Cancer Res. 2020 Apr 15;26(8):1877-1885. doi: 10.1158/1078-0432.CCR-19-3467. Epub 2020 Jan 15. PMID 31941831
- [Background] Caplin ME, Pavel M, Cwikla JB, Phan AT, Raderer M, Sedlackova E, Cadiot G, Wolin EM, Capdevila J, Wall L, Rindi G, Langley A, Martinez S, Blumberg J, Ruszniewski P; CLARINET Investigators. Lanreotide in metastatic enteropancreatic neuroendocrine tumors. N Engl J Med. 2014 Jul 17;371(3):224-33. doi: 10.1056/NEJMoa1316158. PMID 25014687
- [Background] Molina AM, Hu J, Nanus DM. Is Underutilization of Cytoreductive Nephrectomy in Patients With Metastatic Renal Cancer Contributing to Inferior Survival? J Clin Oncol. 2016 Sep 20;34(27):3235-6. doi: 10.1200/JCO.2016.68.4050. Epub 2016 Aug 15. No abstract available. PMID 27528717
- [Background] Ye L, Santarpia L, Gagel RF. The evolving field of tyrosine kinase inhibitors in the treatment of endocrine tumors. Endocr Rev. 2010 Aug;31(4):578-99. doi: 10.1210/er.2009-0031. Epub 2010 Jul 6. PMID 20605972
- [Background] Anand S, Shivashankar R, Kondal D, Garg V, Khandelwal S, Gupta R, Krishnan A, Amarchand R, Poulter N, Reddy KS, Prabhakaran D, Mohan S. Potassium Intake in India: Opportunity for Mitigating Risks of High-Sodium Diets. Am J Prev Med. 2020 Feb;58(2):302-312. doi: 10.1016/j.amepre.2019.09.017. PMID 31959324
- [Background] Fassnacht M, Terzolo M, Allolio B, Baudin E, Haak H, Berruti A, Welin S, Schade-Brittinger C, Lacroix A, Jarzab B, Sorbye H, Torpy DJ, Stepan V, Schteingart DE, Arlt W, Kroiss M, Leboulleux S, Sperone P, Sundin A, Hermsen I, Hahner S, Willenberg HS, Tabarin A, Quinkler M, de la Fouchardiere C, Schlumberger M, Mantero F, Weismann D, Beuschlein F, Gelderblom H, Wilmink H, Sender M, Edgerly M, Kenn W, Fojo T, Muller HH, Skogseid B; FIRM-ACT Study Group. Combination chemotherapy in advanced adrenocortical carcinoma. N Engl J Med. 2012 Jun 7;366(23):2189-97. doi: 10.1056/NEJMoa1200966. Epub 2012 May 2. PMID 22551107
- [Background] Nolan CR, Linas SL. Mechanism of antihypertensive effect of potassium depletion in renovascular hypertension. Am J Physiol. 1988 Nov;255(5 Pt 2):H1181-7. doi: 10.1152/ajpheart.1988.255.5.H1181. PMID 3056041
- [Background] Trotman J, Opat S, Gottlieb D, Simpson D, Marlton P, Cull G, Munoz J, Tedeschi A, Roberts AW, Seymour JF, Atwal SK, Yu Y, Novotny W, Holmgren E, Tan Z, Hilger JD, Huang J, Tam CS. Zanubrutinib for the treatment of patients with Waldenstrom macroglobulinemia: 3 years of follow-up. Blood. 2020 Oct 29;136(18):2027-2037. doi: 10.1182/blood.2020006449. PMID 32698195
- [Background] Ferraro AJ. The Many Fictions of Illness: A Rhetorical Approach to Understanding Fictionality in Mom's Cancer. Lit Med. 2021;39(2):227-248. doi: 10.1353/lm.2021.0022. PMID 34897126
- [Background] REMAP-CAP Investigators; Gordon AC, Mouncey PR, Al-Beidh F, Rowan KM, Nichol AD, Arabi YM, Annane D, Beane A, van Bentum-Puijk W, Berry LR, Bhimani Z, Bonten MJM, Bradbury CA, Brunkhorst FM, Buzgau A, Cheng AC, Detry MA, Duffy EJ, Estcourt LJ, Fitzgerald M, Goossens H, Haniffa R, Higgins AM, Hills TE, Horvat CM, Lamontagne F, Lawler PR, Leavis HL, Linstrum KM, Litton E, Lorenzi E, Marshall JC, Mayr FB, McAuley DF, McGlothlin A, McGuinness SP, McVerry BJ, Montgomery SK, Morpeth SC, Murthy S, Orr K, Parke RL, Parker JC, Patanwala AE, Pettila V, Rademaker E, Santos MS, Saunders CT, Seymour CW, Shankar-Hari M, Sligl WI, Turgeon AF, Turner AM, van de Veerdonk FL, Zarychanski R, Green C, Lewis RJ, Angus DC, McArthur CJ, Berry S, Webb SA, Derde LPG. Interleukin-6 Receptor Antagonists in Critically Ill Patients with Covid-19. N Engl J Med. 2021 Apr 22;384(16):1491-1502. doi: 10.1056/NEJMoa2100433. Epub 2021 Feb 25. PMID 33631065
- [Background] Andre T, Shiu KK, Kim TW, Jensen BV, Jensen LH, Punt C, Smith D, Garcia-Carbonero R, Benavides M, Gibbs P, de la Fouchardiere C, Rivera F, Elez E, Bendell J, Le DT, Yoshino T, Van Cutsem E, Yang P, Farooqui MZH, Marinello P, Diaz LA Jr; KEYNOTE-177 Investigators. Pembrolizumab in Microsatellite-Instability-High Advanced Colorectal Cancer. N Engl J Med. 2020 Dec 3;383(23):2207-2218. doi: 10.1056/NEJMoa2017699. PMID 33264544
- [Background] Ghasemi A, Vaseghi G, Hojjatallah A, Haghjooy Javanmard S. The effects of morphine on vascular cell adhesion molecule 1(VCAM-1) concentration in lung cancer cells. Arch Physiol Biochem. 2023 Apr;129(2):484-488. doi: 10.1080/13813455.2020.1838552. Epub 2021 Jan 15. PMID 33449821
- [Background] Xie N, Shen G, Gao W, Huang Z, Huang C, Fu L. Neoantigens: promising targets for cancer therapy. Signal Transduct Target Ther. 2023 Jan 6;8(1):9. doi: 10.1038/s41392-022-01270-x. PMID 36604431
- [Background] He Y, Lakhani CM, Rasooly D, Manrai AK, Tzoulaki I, Patel CJ. Comparisons of Polyexposure, Polygenic, and Clinical Risk Scores in Risk Prediction of Type 2 Diabetes. Diabetes Care. 2021 Apr;44(4):935-943. doi: 10.2337/dc20-2049. Epub 2021 Feb 9. PMID 33563654
- [Background] Erickson TA, Shih YP, Fass J, Jang M, Tran E. T Cells Engineered to Express Immunoreceptors Targeting the Frequently Expressed Medullary Thyroid Cancer Antigens Calcitonin, CEA, and RET M918T. Thyroid. 2022 Jul;32(7):789-798. doi: 10.1089/thy.2022.0020. PMID 35587601
- [Background] Leidner R, Sanjuan Silva N, Huang H, Sprott D, Zheng C, Shih YP, Leung A, Payne R, Sutcliffe K, Cramer J, Rosenberg SA, Fox BA, Urba WJ, Tran E. Neoantigen T-Cell Receptor Gene Therapy in Pancreatic Cancer. N Engl J Med. 2022 Jun 2;386(22):2112-2119. doi: 10.1056/NEJMoa2119662. PMID 35648703
- [Background] Zheng C, Fass JN, Shih YP, Gunderson AJ, Sanjuan Silva N, Huang H, Bernard BM, Rajamanickam V, Slagel J, Bifulco CB, Piening B, Newell PHA, Hansen PD, Tran E. Transcriptomic profiles of neoantigen-reactive T cells in human gastrointestinal cancers. Cancer Cell. 2022 Apr 11;40(4):410-423.e7. doi: 10.1016/j.ccell.2022.03.005. PMID 35413272
- [Background] Gartner JJ, Parkhurst MR, Gros A, Tran E, Jafferji MS, Copeland A, Hanada KI, Zacharakis N, Lalani A, Krishna S, Sachs A, Prickett TD, Li YF, Florentin M, Kivitz S, Chatmon SC, Rosenberg SA, Robbins PF. A machine learning model for ranking candidate HLA class I neoantigens based on known neoepitopes from multiple human tumor types. Nat Cancer. 2021 May;2(5):563-574. doi: 10.1038/s43018-021-00197-6. Epub 2021 May 3. PMID 34927080
- [Background] Yossef R, Tran E, Deniger DC, Gros A, Pasetto A, Parkhurst MR, Gartner JJ, Prickett TD, Cafri G, Robbins PF, Rosenberg SA. Enhanced detection of neoantigen-reactive T cells targeting unique and shared oncogenes for personalized cancer immunotherapy. JCI Insight. 2018 Oct 4;3(19):e122467. doi: 10.1172/jci.insight.122467. PMID 30282837
- [Background] Nguea P A, Robertson J, Herrera MC, Chymkowitch P, Enserink JM. Desumoylation of RNA polymerase III lies at the core of the Sumo stress response in yeast. J Biol Chem. 2019 Dec 6;294(49):18784-18795. doi: 10.1074/jbc.RA119.009721. Epub 2019 Nov 1. PMID 31676685
- [Background] Orkin J, Major N, Esser K, Parmar A, Couture E, Daboval T, Kieran E, Ly L, O'Brien K, Patel H, Synnes A, Robson K, Barreira L, Smith WL, Rizakos S, Willan AR, Yaskina M, Moretti ME, Ungar WJ, Ballantyne M, Church PT, Cohen E. Coached, Coordinated, Enhanced Neonatal Transition (CCENT): protocol for a multicentre pragmatic randomised controlled trial of transition-to-home support for parents of high-risk infants. BMJ Open. 2021 Jul 7;11(7):e046706. doi: 10.1136/bmjopen-2020-046706. PMID 34233983
- [Background] Oliveira M, Assis DM, Paschoalin T, Miranda A, Ribeiro EB, Juliano MA, Bromme D, Christoffolete MA, Barros NM, Carmona AK. Cysteine cathepsin S processes leptin, inactivating its biological activity. J Endocrinol. 2012 Aug;214(2):217-24. doi: 10.1530/JOE-12-0108. Epub 2012 May 31. PMID 22653842